CLINICAL TRIAL: NCT04108819
Title: Ketogenic Diet for Obesity Hypoventilation Syndrome
Acronym: KETOHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00212924
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Obesity Hypoventilation Syndrome; Ketogenic Dieting; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Respiratory Insufficiency | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Experimental): Participants will receive the ketogenic diet.
  Interventions: Dietary Supplement: Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — Subjects will undergo ketogenic diet at a 2.5:1 (fat: carb + protein) ratio for a 2-week period.

SUMMARY:
Obesity hypoventilation syndrome (OHS) is a condition that occurs in small percentage of obese people that causes high carbon dioxide and low oxygen levels in the blood. OHS is associated with respiratory failure, pulmonary hypertension, and death. The cause of OHS is unclear. Since not all obese people develop OHS, it is believed that hormone imbalances can contribute to the breathing problem.

Some diets can change the body's hormones. For example, low-carbohydrate, high fat "ketogenic" diets (KD) may decrease insulin and glucose levels and increase sensitivity to other hormones. The investigators hypothesize that a KD will improve breathing in OHS patients, even in the absence of weight loss.

DETAILED DESCRIPTION:
Obesity hypoventilation syndrome (OHS) is a condition that occurs in small percentage of obese people, that leads to high carbon dioxide levels and low oxygen levels in the blood. OHS is associated with respiratory failure, pulmonary hypertension, hospital admissions, and death. Unfortunately, there is no treatment for OHS besides massive weight loss which often requires bariatric surgery.

In this study, the investigators are examining whether switching from a regular diet to a ketogenic diet will improve breathing, oxygen, and carbon dioxide levels in OHS patients. After a few days-weeks on KD, hormone changes are known to occur and the investigators are examining whether these hormonal changes could stimulate breathing.

This is a pilot study to examine the effects of a 12 day KD on OHS. The outcomes of the study include blood oxygen, carbon dioxide levels, plasma levels of hormones such as insulin, leptin, sleep studies, body composition a, weight, and metabolic rate.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI≥30 kg/m2)
* Hypercapnia (PaCO2>45 or PvCO2>50) on blood gas, OR a sleep study with end-tidal/transcutaneous CO2 monitoring showing an awake CO2 level >50
* Participants without blood gas data may also have suspected OHS on the basis of serum bicarbonate >=28 mEq/L
* Lack of an alternative pulmonary diagnosis that adequately explains hypercapnia. Note that a documented pulmonary diagnosis (e.g. chronic obstructive pulmonary disease (COPD) or asthma) per se will not necessarily exclude subjects, since OHS is often misdiagnosed as obstructive lung disease. Functional or radiographic data must corroborate the presence of the alternate diagnosis.
* Subjects must have had a sleep study and clinical evaluation for sleep apnea. Most subjects with OHS are expected to have concomitant obstructive sleep apnea (OSA). This information is necessary to determine whether continuous positive airway pressure (CPAP)/noninvasive ventilation (NIV) will be used on the research sleep studies.

Exclusion Criteria:

* Concomitant participation in another weight loss or diet program
* Patients with diabetes taking Sodium-glucose Cotransporter-2 (SGLT2) inhibitors (due to risk of diabetic ketoacidosis)
* Patients with type 1 diabetes
* Any patients with a history of diabetic ketoacidosis
* Patients with incomplete sleep apnea diagnosis or management (i.e. those still acclimating to CPAP, or pending therapeutic decisions about OSA management)
* Known or suspected abuse of narcotics or alcohol
* Liver cirrhosis
* Uncontrolled gout
* History of chronic renal insufficiency requiring dialysis
* Females who are pregnant, breast-feeding, or intending to become pregnant
* Food allergies or diet restrictions that research nutritionists cannot accommodate

FOLLOW THIS LINK TO SEE IF YOU QUALIFY:

https://mrprcbcw.hosts.jhmi.edu/redcap/surveys/?s=RYX7DELK9Y

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Change in Awake venous carbon dioxide (PvCO2) Level | Baseline (pre keto diet) and 2 weeks post keto diet
  Measured in mmHg.

SECONDARY OUTCOMES:
Change in Venous pH | Once per week, over 4 weeks
  Measured in moles per liter.
Change in Glucose level | Once per week, over 4 weeks
  Measured in g/dL.
Change in Insulin level | Once per week, over 4 weeks
  Measured in mIU/L.
Change in leptin level | Once per week, over 4 weeks
  Measured in ng/mL.
Change in beta-Hydroxybutyrate level | Once per week, over 4 weeks
  Measured in mg/dL.
Glucose profile | Continuously measured over 4 weeks
  Using continuous glucose monitoring (CGM), to measured glucose level (g/dL) each day at home.
Change in Body weight (kg) | Once per week, over 4 weeks
Change in Oxygen saturation | Once per week, over 4 weeks
  Measured as a percentage.
Change in Blood Pressure | Once per week, over 4 weeks
  Measured in mmHg.
Change in percentage of body fat | Once every 2 weeks, over 4 weeks
  The investigators will measure percentage body fat using the Bioelectrical impedance analysis (BIA).
Change in Apnea Hypopnea Index | Once every 2 weeks, over 4 weeks
  The apnea hypopnea index (AHI) is derived from combined information from EEG signals, flow sensors, respiratory belts, and carbon dioxide censors and is a measure of severity of sleep apnea. AHI < 5 is considered normal. AHI 5-15 is considered mild sleep apnea. AHI 15-30 is considered moderate sleep apnea. AHI >30 is considered severe sleep apnea.
Change in LDL Cholesterol | Once per week, over 4 weeks
  Measured in mg/dL.
Change in HDL Cholesterol | Once per week, over 4 weeks
  Measured in mg/dL.
Change in Triglyceride level | Once per week, over 4 weeks
  Measured in mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States